CLINICAL TRIAL: NCT04166045
Title: Evaluation of Peripheral Nerve Stimulation for Acute Treatment of Migraine Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theranova, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CRD-01-1282-01
Record Dates: First submitted 2019-11-13; First posted 2019-11-18 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Episodic Migraine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham (Sham Comparator): Treatment at the bicep location
  Interventions: Device: Sham Treatment Location
- Verum (Active Comparator): Treatment at the hand location
  Interventions: Device: Verum Treatment Location

INTERVENTIONS:
Device: Sham Treatment Location — The device applies transcutaneous electrical nerve stimulation to the bicep
  Arms: Sham
Device: Verum Treatment Location — The device applies transcutaneous electrical nerve stimulation to the hand
  Arms: Verum

SUMMARY:
Clinical study to determine the responder rate of the TheraNova Migraine Treatment System to that of a sham control treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18-100 years, inclusive
* Diagnosis of episodic migraine with and without aura per International Headache Society diagnostic criteria
* 4-14 migraine days per month
* Ability to provide informed consent
* Demonstrates no contraindication to the use of electrical nerve stimulation
* Capable and willing to follow all study-related procedures

Exclusion Criteria:

* Currently pregnant or breastfeeding, pregnant within the past 6 months or intends to become pregnant during the enrollment period
* Diagnosis of chronic migraine or other forms of primary or secondary headache disorders, including medication overuse headache per International Headache Society diagnostic criteria
* Any medical condition that would, in the opinion of the investigator, make the subject ineligible
* Has received botulinum toxin injections within the past 3 months
* Is currently implanted with an electrical and/or neurostimulator devic, including but not limited to cardiac pacemaker or defibrillator, vagal neurostimulator, sacral stimulator, bone growth stimulator, or cochlear implant
* Use of investigational drug/device therapy within the past 4 weeks
* Deemed unsuitable for enrollment in study by the investigator based on subjects' history or physical examination (including bleeding disorders, anticoagulant medications and peripheral neuropathy)
* No changes in preventive medications (or other medications determined to potentially interfere with the study) in the previous 30 days and no intent to change it during the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-04-29 (Actual)

PRIMARY OUTCOMES:
Mean change in pain score | 4 months
  We will also assess the change in migraine pain before versus after treatment with the 100-mm Visual Analogue Scale (VAS), which is a continuum scale that patients can quantify their pain from none (0 mm) to extreme (100 mm) for both treatment sites. The mean score for each patient cohort will be calculated. We will also perform a sub analysis on women versus men.
Percent of subjects who are responders | 4 months
  For each subject treatment effectiveness will be assessed by both achieving pain relief (if the pain decreases from a 4-point visual rating scale (VRS) of 'severe' or 'moderate' at pre-treatment to 'mild' or 'none' at 120-min post-treatment) or pain-free ('none') status. The percent of subjects that experience a significant reduction in pain relief score (VRS) will be calculated for the verum and sham treatment sites.

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Scottsdale, Arizona, United States